CLINICAL TRIAL: NCT00260130
Title: Study 1: Viscosity Study Study 2: Meal Timing Study Study 3:Chronic Fluid and Solid Food Intake in Lean and Overweight Individuals
Brief Title: Food Rheology and Feeding in Lean and Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Mattes, Prof. Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DK63185 (completed); R01DK063185 (NIH); Study 1: 503001275; Study 2: 508002908; Study 3: 505002589
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Overweight; Diabetes
Keywords: obesity; food intake; human; energy balance; beverage
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus | interventions — Food

ARMS (2):
- 1 (Active Comparator): Consuming fruit and vegetable juice
  Interventions: Other: food in fluid form
- 2 (Active Comparator): Consuming whole fruits and vegetables
  Interventions: Other: food in solid form

INTERVENTIONS:
Other: food in fluid form — dietary intake of fluid forms of vegetables
  Arms: 1
Other: food in solid form — dietary intake of solid forms of vegetables
  Arms: 2

SUMMARY:
The 2010 National Health Objectives call for a reduction in the prevalence of obesity. The marked recent increase in overweight and obesity prevalence implicates behavioral factors in the etiology of the epidemic. The present proposal hypothesizes the trend is attributal, in part, to increasing consumption of energy-yeilding beverages since they are a significant and increasing source of dietarty energy and they elicit weaker appetitive and dietary responses than solid foods.

DETAILED DESCRIPTION:
Three human studies are propsed to more fully characterized attributes of liquids and solids that may account for the differential appetitive responses they elicit, potential contributory mechanisms as well as the dietary implications of their consumption. Study 1 will contrast the acute effects of fluid and solid foods varying in macronutrient content on satiation, satiety and feeding. Study 2 will determine if the pattern of fluid and solid ingestion influences satiety and feeding by monitoring appetitive and dietary responses to energy and macronutrient matched fluid and solid loads ingested as meal components or between meal snacks. To better assess the clinical implications ofdiets incorpprating liquid or solid supplements. Study 3 will entail chronic ingestion of matched energy yeilding fluid or solid loads with concurrent measurement of appetite, dietary intake, energy expenditureand body weight/composition.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-23 or 27-35
* weight stable
* constant habitual activity pattern
* low fruit/vegetable consumer
* non-restrained eater

Exclusion Criteria:

* diabetic
* taking medication known to influence appetite

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
satiation and satiety on liquid verses solid foods with concurrent measurements of appetite, dietary intake, energy expenditure and body weight/composition. | 8 weeks

SECONDARY OUTCOMES:
cephalic phase testing at week 8 | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, MPH, PhD, RD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- See also: Dr. Mattes Laboratory for Sensory and Ingestive Studies web site. — http://www.foodsci.purdue.edu/research/27